CLINICAL TRIAL: NCT07209397
Title: A Randomized, Prospective, Multicenter, Double-Blind, Sham-Controlled Study to Assess the MORPHEUSV Radiofrequency (RF) Device in the Treatment of Female Patients With Idiopathic Overactive Bladder (OAB) With Urge Incontinence and/or Urge-Predominant Mixed Incontinence
Brief Title: Detrusor Nerve Radiofrequency Ablation for Overactive Bladder in Women
Acronym: DENARA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Collaborators: Foundation for Female Health Awareness (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DO614953A
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-08

CONDITIONS: Overactive Bladder; Overactive Bladder (OAB); Urge Urinary Incontinence; Mixed Urinary Incontinence (Urge-Predominant); Mixed Urinary Incontinence; Idiopathic Overactive Bladder With Urinary Incontinence; Idiopathic Overactive Bladder
Keywords: Overactive bladder; Urge urinary incontinence; Mixed urinary incontinence; Female urinary symptoms; urogynecology; Female Urology
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to receive either a single session of the MORPHEUS V radiofrequency (RF) treatment or a sham procedure. The study uses a parallel assignment model in which participants remain in their assigned group through the 6-month primary endpoint. After completing the 6-month visit, participants in the sham group may elect to cross over and receive the active treatment. All participants will be followed for 12 months from the time of their initial intervention to assess safety and durability of treatment effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- MORPHEUSV Treatment Arm (Active Comparator): Participants in this arm will receive a single session of radiofrequency (RF) treatment using the MORPHEUSV device. The treatment is delivered vaginally using a bipolar RF applicator at a therapeutic energy setting. No anesthesia is required. Participants will be followed for 12 months to evaluate safety and effectiveness.
  Interventions: Device: Detrusor nerve radiofrequency ablation
- Sham Control Arm (Sham Comparator): Participants in this arm will undergo a procedure using a visually identical MORPHEUSV applicator, but without RF energy delivery (sham). The procedure mimics the appearance and duration of the active treatment. Participants will be followed for 12 months. After completing the 6-month follow-up, they may elect to cross over and receive a single session of the active RF treatment.
  Interventions: Device: Simulated (sham) detrusor nerve radiofrequency ablation

INTERVENTIONS:
Device: Detrusor nerve radiofrequency ablation — A single, vaginal radiofrequency (RF) treatment. The procedure is performed with a bipolar RF applicator and requires no anesthesia. Delivered in a single session in an outpatient setting.
  Arms: MORPHEUSV Treatment Arm
Device: Simulated (sham) detrusor nerve radiofrequency ablation — A simulated (sham) radiofrequency (RF) treatment, but with no energy delivered. The procedure mimics the appearance, duration, and positioning of the active device, without therapeutic effect.
  Arms: Sham Control Arm

SUMMARY:
The goal of this clinical trial is to learn if a vaginal radiofrequency (RF) device called MORPHEUSV works to treat overactive bladder (OAB) in women. Researchers also want to learn how safe the device is for this indication. This study will include women ages 22 to 80 who have had OAB symptoms for at least 6 months. The main questions it aims to answer are: Does the MORPHEUSV device lower the number of daily episodes of accidental urine leakage caused by urgency? Does it work better than a sham (placebo) treatment? Researchers will compare the MORPHEUSV device to a sham treatment to see how well it reduces symptoms of overactive bladder. Participants will: 1) Receive one session of either the MORPHEUSV or sham treatment. 2) Track their symptoms using a diary and questionnaires 3) Return for three to six follow-up visits over 12 months. This study is being conducted at multiple clinics in the United States.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a common condition that significantly impacts the quality of life in women, especially those with urge urinary incontinence (UUI) or mixed incontinence with a predominant urgency component. Current treatments for OAB, including behavioral therapy and pharmacologic agents, often have limited long-term efficacy, tolerability issues, or low adherence rates. There is a significant need for alternative, non-invasive therapies that can provide symptom relief with fewer side effects. The MORPHEUSV system is a vaginally delivered radiofrequency (RF) energy device designed to remodel submucosal tissue through controlled thermal stimulation. This technology is currently being investigated for its ability to improve bladder control by targeting pelvic tissue support and neuromodulation pathways. The device is investigational for this indication and is being studied under an FDA-approved Investigational Device Exemption (IDE G250071). This is a prospective, randomized, multicenter, double-blind, sham-controlled clinical trial designed to evaluate the safety and efficacy of the MORPHEUSV RF device in women aged 22 to 80 with idiopathic OAB and at least 7 episodes of UUI per week. The study will enroll approximately 202 participants at up to 12 sites across the United States. Participants will be randomized 2:1 to either a single session of active RF treatment or a sham (placebo) treatment. The primary outcome is the proportion of participants achieving a ≥50% reduction in UUI episodes from baseline at 6 months. Secondary and exploratory outcomes include symptom reduction across urgency, frequency, nocturia, and quality of life metrics, as well as device-related adverse events. Blinding will be maintained through the use of an identical sham applicator with no RF energy delivery. A crossover option is available for sham subjects who complete the 6-month follow-up, allowing them to receive the active treatment. All participants will be followed for 12 months after their initial intervention to evaluate durability of response and long-term safety. An internal data review committee will periodically evaluate cumulative safety data. The study is conducted under Good Clinical Practice (GCP) guidelines and will be overseen by Sterling IRB.

ELIGIBILITY:
INCLUSION CRITERIA:

* Female, aged 22 to 80 years inclusive at the time of consent.
* History of idiopathic overactive bladder (OAB) symptoms for ≥6 months.
* At least 7 episodes of urge urinary incontinence (UUI) over 3 days, as recorded in a 3-day bladder diary during screening.
* Urge-predominant incontinence, defined as greater number of UUI episodes than stress urinary incontinence (SUI) episodes during screening.
* Willing and able to complete the 3-day bladder diary.
* Willing to discontinue OAB medications (e.g., anticholinergics, beta-3 agonists) at least 2 weeks prior to baseline treatment visit, if currently taking such medications.
* Willing to use a reliable method of contraception during the study period, if of childbearing potential and sexually active.
* Negative pregnancy test at screening (if applicable).
* Willing and able to provide written informed consent and comply with study procedures and follow-up schedule.

EXCLUSION CRITERIA:

* Predominant stress urinary incontinence (SUI) based on bladder diary
* Currently pregnant, breastfeeding, or planning pregnancy during the study
* History of neurologic conditions affecting bladder function (e.g., multiple sclerosis, spinal cord injury, Parkinson's disease)
* Active urinary tract infection (UTI) at screening
* History of interstitial cystitis, bladder pain syndrome, or chronic pelvic pain
* Prior or current bladder cancer, pelvic malignancy, or pelvic radiation
* Pelvic organ prolapse beyond the hymen (POP-Q stage > II)
* Implanted neuromodulation device or prior sacral nerve stimulation
* Use of bulking agents, Botox, or surgical treatment for incontinence within 12 months
* Prior pelvic floor RF treatment or laser vaginal rejuvenation
* Significant pelvic anatomical abnormalities that interfere with treatment
* Use of investigational drug or device within 30 days before screening
* Any condition that, in the investigator's opinion, would interfere with safe study participation or data integrity
* Uncontrolled systemic disease (e.g., uncontrolled diabetes, cardiovascular disease)
* Inability or unwillingness to comply with study requirements or follow-up

Ages: 22 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving ≥50% reduction in weekly urge urinary incontinence (UUI) episodes | 6 months post-treatment
  The percentage of participants who achieve at least a 50% reduction from baseline in the number of UUI episodes per week, as recorded in a 7-day bladder diary. This is the primary efficacy endpoint used to evaluate the effectiveness of the MORPHEUSV device compared to sham.

SECONDARY OUTCOMES:
Change from baseline in mean number of UUI episodes per week | 6 months
  Mean change in UUI episodes per week from baseline, based on 7-day bladder diary.
Change from baseline in mean number of urgency episodes per week | 6 months
  Mean change in urgency episodes per week from baseline, based on bladder diary.
Change from baseline in mean number of micturitions per 24 hours | 6 Months
  Change in average number of daily voids as measured via bladder diary.
Change from baseline in Incontinence Quality of Life (I-QOL) total score | 6 Months
  Mean change from baseline in total score on the Incontinence Quality of Life Questionnaire (I-QOL), a validated 22-item patient-reported outcome measure assessing the impact of urinary incontinence on quality of life. Total scores range from 0 to 100, with higher scores indicating better quality of life.
Change from baseline in Urgency Perception Scale (UPS) score | 6 Months
  Mean change from baseline in urgency perception severity measured using the Urgency Perception Scale (UPS), a validated patient-reported scale assessing urinary urgency severity. UPS scores range from 0 to 3, with higher scores indicating greater urgency severity (worse symptoms).
Incidence and severity of adverse events | 12 Months
  Frequency and severity of treatment-emergent adverse events in each arm, collected at all follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mickey Karram, MD, Study Director — Foundation for Female Health Awareness (FFHA)
Locations (9):
- United States (9):
  - Stanford Medicine Department of Obstetrics & Gynecology, Palo Alto, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Advanced Specialty Research, Boise, Idaho
  - University of Chicago Medicine Urogynecology, Chicago, Illinois
  - Cypress Medical Research Center, Wichita, Kansas
  - Bay State Clinical Trials, Watertown, Massachusetts
  - Urology Center, P.C., Omaha, Nebraska
  - UNLV Kirk Kerkorian School of Medicine Department of Gynecologic Surgery & Obstetrics, Las Vegas, Nevada
  - Atrium Health Wake Forest Female Pelvic Health Division, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided